CLINICAL TRIAL: NCT03245749
Title: Effect of Oily Fish Intake, Sex, Age, BMI, and APOE Genotype on Plasma Long Chain n-3 Fatty Acid Composition
Status: Completed | Type: Observational
Sponsor: University of Southampton (Other)
Collaborators: Food Standards Agency, United Kingdom (Other Government); Ocean Nutrition (Industry)
Responsible Party: Sponsor
Other Study IDs: RRD7/N02/A
Record Dates: First submitted 2017-08-07; First posted 2017-08-10 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Plasma Omega-3 Status
Keywords: omega-3 status; blood lipids; Eicosapentaenoic acid (EPA); Docosahexaenoic acid (DHA)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood and plasma samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this study is to investigate the effect of habitual oily fish intake, sex, age, BMI, and APOE genotype on plasma long chain n-3 fatty acid composition.

DETAILED DESCRIPTION:
The marine long chain n-3 polyunsaturated fatty acids (LC n-3 PUFAs) eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA) are beneficial to cardiovascular and cognitive health and the concentration of EPA and DHA present in blood and tissue lipids is positively correlated with these effects.

As a result, national and global authorities recommend regular consumption of oily fish in order to provide approximately 500 mg EPA+DHA per day in a healthy population. However, the associations between EPA and DHA intake and blood and tissue status, and therefore physiological benefits, are highly variable and the factors influencing this heterogeneity are not well understood.

This study aims to investigate the effect of habitual oily fish intake as well as sex, age, BMI, and Apolipoprotein E (APOE) genotype on LC n-3 PUFA status in plasma phosphatidylcholine, non-esterified fatty acids, cholesteryl esters and triacylglycerols in order to obtain greater knowledge of the determinants of LC n-3 PUFA status with the potential to develop more robust, and perhaps subgroup specific, recommendations for EPA and DHA intake.

ELIGIBILITY:
Exclusion Criteria:

* Diagnosed endocrine dysfunction including diabetes
* Fasting glucose concentration > 6.5 mmol/L
* Myocardial infarction in the previous 2 years
* The use of medication that may interfere with lipid metabolism
* Fasting total cholesterol of > 8.0 mmol/L
* TG of > 3.0 mmol/L
* Currently following a weight loss diet
* Taking n-3 fatty acid supplements

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Individuals residing in Southampton, East Anglia, Glasgow and Newcastle
Sampling Method: Probability Sample
Enrollment: 374 (Actual)
Dates: Start 2003-06 (Actual); Primary Completion 2005-09 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Plasma long chain n-3 polyunsaturated fatty acid concentrations | Baseline
  Concentrations of eicosapentaenoic acid (EPA), docosapentaenoic acid (DPA) and docosahexaenoic acid (DHA) in plasma phosphatidylcholine, non-esterified fatty acids, cholesteryl esters and triacylglycerols

SECONDARY OUTCOMES:
APOE genotyping | Baseline
  APOE genotype determined from blood sample
Anthropometric measurements | Baseline
  Height and weight to determine BMI

CONTACTS AND LOCATIONS:
Overall Officials: Philip C Calder, Principal Investigator — University of Southampton
Locations (5):
- United Kingdom (5):
  - University of Glasgow, Glasgow
  - Newcastle University, Newcastle upon Tyne
  - Univeristy of East Anglia, Norwich
  - University of Reading, Reading
  - University of Southampton, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fisk HL, Irvine M, Miles EA, Lietz G, Mathers JC, Packard CJ, Armah CK, Kofler BM, Curtis PJ, Minihane AM, Calder PC. Association of oily fish intake, sex, age, BMI and APOE genotype with plasma long-chain n-3 fatty acid composition. Br J Nutr. 2018 Jul;120(1):23-32. doi: 10.1017/S000711451800106X. Epub 2018 May 6. PMID 29729672